CLINICAL TRIAL: NCT00699023
Title: Effects of Ezetimibe in Association With Statins on Postprandial Lipemia in Type 2 Diabetic Patients
Brief Title: Ezetimibe and Statins on Postprandial Lipemia in Type 2 Diabetes
Acronym: EZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Angela A. Rivellese, MD, Department of Clinical and Experimental Medicine Federico II University Naples
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 239/07
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: Postprandial Lipemia; Type 2 Diabetes
Keywords: postprandial lipemia; type 2 diabetes; ezetimibe; hypercholesterolemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): ezetimibe tablets 10 mg/die + simvastatin tablets 20 mg/die six weeks
  Interventions: Drug: ezetimibe tablets; Drug: simvastatin tablets
- 2 (Placebo Comparator): placebo + simvastatin tablets 20 mg/die six weeks
  Interventions: Drug: simvastatin tablets; Drug: placebo

INTERVENTIONS:
Drug: ezetimibe tablets — ezetimibe tablets 10 mg/die
  Arms: 1
Drug: simvastatin tablets — simvastatin tablets 20 mg/die
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether ezetimibe in association with statins is more effective than statins alone on postprandial lipemia in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes since at least two years
* Stable metabolic control (HbA1c<8.0%) for at least six months on diet or diet+oral hypoglycemic drugs (insulin secretagogues or metformin), not to be changed during the study period.
* BMI<30 kg/m2 and body weight stable during the last six months.
* Both sexes; only post-menopausal women.
* LDL-cholesterol >130 mg/dl, plasma triglycerides <400 mg/dl.
* No use of hypolipidemic drugs in the last three months.

Exclusion Criteria:

* Patient with renal (serum creatinine >1.5 mg/dl) or hepatic (serum transaminases >three times upper normal values) impairment.
* Patients with history of cardiovascular disease.
* Pre-menopausal women.
* Any other acute or chronic degenerative disease.
* Anemia (Hb<12 g/dl).
* Uncontrolled blood pressure.
* Use of any drugs able to interfere with the study medications

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Incremental AUC after a fat-rich meal of cholesterol concentration in chylomicron and VLDL fractions | 6 weeks

SECONDARY OUTCOMES:
Incremental AUC after a fat rich-meal of apo B48 concentration- marker of the number of intestinally derived lipoproteins- in chylomicron and VLDL | 6 weeks
Fasting LDL concentration | 6 weeks
Cholesterol/triglyceride ratio in postprandial chylomicrons and VLDL fractions. | 6 weeks
Postprandial LDL size | 6 weeks
Concentration and Composition of different lipoprotein subclasses in the fasting condition. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Riccardi, Prof, Study Chair — Department of Clinical and Experimental Medicine, Federico II University Hospital, Naples, Italy
Locations (1):
- Department of Clinical and Experimental Medicine, Federico II University Hospital,, Naples, Naples, Italy

REFERENCES:
- [Background] Rivellese AA, De Natale C, Di Marino L, Patti L, Iovine C, Coppola S, Del Prato S, Riccardi G, Annuzzi G. Exogenous and endogenous postprandial lipid abnormalities in type 2 diabetic patients with optimal blood glucose control and optimal fasting triglyceride levels. J Clin Endocrinol Metab. 2004 May;89(5):2153-9. doi: 10.1210/jc.2003-031764. PMID 15126535
- [Background] Annuzzi G, De Natale C, Iovine C, Patti L, Di Marino L, Coppola S, Del Prato S, Riccardi G, Rivellese AA. Insulin resistance is independently associated with postprandial alterations of triglyceride-rich lipoproteins in type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2004 Dec;24(12):2397-402. doi: 10.1161/01.ATV.0000146267.71816.30. Epub 2004 Sep 30. PMID 15458975
- [Background] Davidson MH, Toth PP. Combination therapy in the management of complex dyslipidemias. Curr Opin Lipidol. 2004 Aug;15(4):423-31. doi: 10.1097/01.mol.0000137221.16160.b9. PMID 15243215